CLINICAL TRIAL: NCT05590572
Title: A Study of Etoposide and Ifosfamide Combined With or Without Sulfatinib on Relapsed or Refractory Drug Resistant Osteosarcoma
Brief Title: A Study of Sulfatinib on Relapsed or Refractory Drug Resistant Osteosarcoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Chonnam National University (Other); Peking University People's Hospital (Other); Qilu Hospital of Shandong University (Other); Ruijin Hospital (Other); Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-0880
Record Dates: First submitted 2022-10-19; First posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Osteosarcoma
Keywords: Refractory or Relapsed osteosarcoma; Sulfatinib; Tyrosine kinase inhibitors; Etoposide; Ifosfamide
MeSH Terms: conditions — Osteosarcoma | interventions — surufatinib; Etoposide; Ifosfamide

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Etoposide plus Ifosfamide group (Active Comparator): Children and adolescents with relapsed or refractory drug resistant osteosarcoma
  Interventions: Drug: Etoposide; Drug: Isophosphamide
- Etoposide plus Ifosfamide Combined With Sulfatinib (Experimental): Children and adolescents with relapsed or refractory drug resistant osteosarcoma
  Interventions: Drug: Sulfatinib; Drug: Etoposide; Drug: Isophosphamide

INTERVENTIONS:
Drug: Sulfatinib — (1) Sulfatinib: 300 mg, oral once a day (QD), 21 days as a cycle
  Arms: Etoposide plus Ifosfamide Combined With Sulfatinib
Drug: Etoposide — (1) Etoposide: 100 mg/m2/day (initial dose) will be administered on the first to third days of each 21 day cycle, a total of 5 cycles. The dose of etoposide can be reduced to 80 mg/m2/day and 60 mg/m2/day.;
Drug: Isophosphamide — (1) Isophosphamide: 3000 mg/m2/day (initial dose) will be administered on the first to third days of each 21 day cycle for 5 cycles. The dose of ifosfamide can be reduced to 2400 mg/m2/day and 1800 mg/m2/day.

SUMMARY:
This is a phase 1/2 study evaluating safety, tolerability, and efficacy of Sulfatinib in combination with chemotherapy (ifosfamide and etoposide) in children and adolescents with refractory or relapsed osteosarcoma ( combination Sulfatinib).

DETAILED DESCRIPTION:
The study consists of 2 cohorts:

Cohort 1 (Traditional chemotherapy) will evaluate the efficacy of ifosfamide and etoposide in children, adolescents, and young adults with relapsed or refractory osteosarcoma.

Cohort 2 (Combination Expansion) will evaluate the efficacy of Sulfatinib in combination with ifosfamide and etoposide in children, adolescents, and young adults with relapsed or refractory osteosarcoma.

Sulfatinib will be provided as hard capsules containing 300 mg Sulfatinib. Sulfatinib capsules should be dissolved in water or apple juice for those who are unable to swallow capsules.

ELIGIBILITY:
Inclusion Criteria:

1. Osteosarcoma subjects Male or female participants aged 2 to 25 years at the time of informed consent(Histologically or cytologically confirmed diagnosis of high grade osteosarcoma)
2. Recurrent or refractory solid tumor malignancies that have treated with standard anticancer therapy but have no available treatment options.
3. Evaluable or measurable disease that met the following criteria: 1. Participants must have an evaluable or measurable disease based on RECIST 1.1, using computed tomography (CT)/ magnetic resonance imaging (MRI). 2. Lesions that have been treated locally, such as external beam radiation therapy (EBRT) or radiofrequency (RF) ablation, must subsequently grow clearly to be considered target lesions.
4. Life expectancy is 3 months or more.
5. Adequate bone marrow function : ①. Absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L. ②. Hemoglobin ≥ 8.0 g/ deciliter (hemoglobin ≤ 8.0 g/ deciliter is acceptable if corrected by growth factors or transfusion before starting sovanitinib). ③. Platelet count ≥ 75 x 10^9/L.
6. Adequate liver function: 1. Bilirubin ≤ 1.5 times the upper limit of normal (ULN). 2. Alkaline phosphatase, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 times of ULN.
7. Adequate renal function, such as creatinine clearance (or radioisotope glomerular filtration rate [GFR]), must be greater than 70 mL/min/ 1.73 square meters.

(8)A baseline left ventricular ejection fraction (LVEF) of 50% or greater, as determined by echocardiography, indicates adequate cardiac function.

(9) Good control of blood pressure (BP) with or without antihypertensive medication was defined as : blood pressure below 95% for sex, age, and height/length at screening (according to National Heart, Lung, and Blood Institute guidelines) and no change in antihypertensive medication during the cycle 1 of project. participants with osteosarcoma had blood pressure ≤150/90 mm Hg at screening and had no change in antihypertensive therapy during the cycle 1 of project.

(10)Parents or legal representative (guardian) shall sign the written informed consent and obtain the consent of minor participants. Written informed consent from subjects ≥18 years of age. Willing and able to abide by the researchers determine solutions, plans, and toxicity of follow-up management.

Exclusion Criteria:

1. Any active infection or infectious disease.
2. Any medical condition or other condition that the investigator believes will prevent the participant from participating in the clinical study.
3. Other organ toxicity (except hair loss) caused by previous anti-cancer treatment (research drug, chemotherapy or radiotherapy)
4. Known hypersensitivity to any component of the product (soventinib or ingredient).
5. Any other anti-tumor treatment is given at the same time.
6. He has been treated with sovantinib before.
7. Two or more previous VEGF/VEGFR targeted therapies.
8. Currently receiving any study drug or device in another clinical trial or within 30 days before informed consent.
9. Clinically significant ECG abnormalities, including significant baseline QT or QTc interval prolongation (e.g., QTc interval duplication is demonstrated to be greater than 480 milliseconds).
10. Gastrointestinal malabsorption or any other condition that the investigator believes may affect the absorption of sovantinib.
11. Gastrointestinal bleeding or active hemoptysis (at least half a teaspoon of bright red blood) occurred within 3 weeks before the first administration of the study drug.
12. Active second malignant tumor (excluding superficial melanoma, in situ, basal or squamous cell skin cancer with definite treatment) within 2 years before enrollment.
13. Previously treated with ifosfamide with nephrotoxicity or encephalopathy grade greater than or equal to grade 3.

Women who were breastfeeding or pregnant at the time of screening or baseline. If a negative screening pregnancy test is obtained more than 72 hours before the first administration of the study drug, a separate baseline assessment is required.

-

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 148 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
4 months progression-free survival | 4 months
  The proportion of patients who had no objective tumor progression or death from the start of treatment to 4 months of follow-up.
Efficacy evaluation in solid tumors | 2 months
  Complete response (CR), all target and non-target lesions (non-lymph nodes) disappear, and the diameter of all pathologic lymph nodes (both target and non-target) must be reduced to <10 mm; Partial response (PR), using baseline total diameter as reference, reduced the total diameter of target lesions by at least 30%.

SECONDARY OUTCOMES:
Best of response,BOR | 4 months
  From the date of the first administration of the study drug to disease progression or death, whichever occurs first.
Duration of Remission (DOR) | 2 years
  Complete response (CR)/ partial response (PR) was first recorded until disease progression was first recorded until the data cutoff date.

CONTACTS AND LOCATIONS:
Overall Officials: zhaoming Ye, PhD, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University; Binhao Li, PhD, Study Director — Second Affiliated Hospital, School of Medicine, Zhejiang University; zengjie zhang, MD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University; Shengdong Wang, MD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University; Xin Huang, PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University; Peng Lin, MD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (5):
- China (4):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Department of Orthopaedic Surgery, Sixth People's Hospital, Shanghai Jiao Tong University,, Shanghai, Shanghai Municipality
- Department of Orthopedic Surgery Chonnam National University, Donggu, Gwangju, South Korea

IPD SHARING:
Plan to Share IPD: No